CLINICAL TRIAL: NCT05765071
Title: Treatment of Lower Leg Anterolateral Chronic Exertional Compartment Syndrome With Intra-muscular Botulinum Injections.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Calgary (Other)
Collaborators: Canadian Academy of Sport and Exercise Medicine (CASEM) (Unknown); Kinesis Medical Centre Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REB22-0439
Record Dates: First submitted 2023-02-15; First posted 2023-03-13 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-02

CONDITIONS: Chronic Exertional Compartment Syndrome
Keywords: anterolateral; CECS; lower leg
MeSH Terms: conditions — Chronic Exertional Compartment Syndrome | interventions — Botulinum Toxins, Type A; Saline Solution

STUDY DESIGN:
Intervention Model Description: Participants receiving botulinum toxin will be compared to those receiving normal saline.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be blinded to the treatment they received until after the 24-week visit is completed. The physiatrist administering the injection and the physiatrist performing the manual muscle power assessments will be blinded to treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Active Comparator): Botulinum toxin (Botox) injection
  Interventions: Biological: Botulinum toxin A
- Control (Placebo Comparator): Normal saline injection
  Interventions: Biological: Normal saline

INTERVENTIONS:
Biological: Botulinum toxin A — Botulinum injections will be prepared by diluting 100 units of botulinum toxin A with 5.0mL of saline (20.0U/mL). A total of 100 units (5.0mL) of botulinum toxin A will be injected into the tibialis anterior, peroneus longus and peroneus brevis muscles of the affected leg. Under ultrasound guidance, the injectant will be deposited at two sites in each muscle near the motor points.
  Other Names: Botox
  Arms: Treatment
Biological: Normal saline — A total of 5.0mL of normal saline will be injected into the tibialis anterior, peroneus longus and peroneus brevis muscles of the affected leg. Under ultrasound guidance, the injectant will be deposited at two sites in each muscle near the motor points.
  Other Names: Placebo
  Arms: Control

SUMMARY:
The goal of this pilot triple-blind randomized clinical trial is to determine the effectiveness of intra-muscular botulism injection for treatment of lower leg anterolateral chronic exertional compartment syndrome (CECS).

Primary Research Question: What is the effectiveness of intra-muscular botulinum injection, compared to normal saline placebo, for reducing pain related to painful sport activity in patients with lower leg anterolateral chronic exertional compartment syndrome (CECS), over a 24-week period?

Secondary outcomes will measure the time to initial onset and duration of pain during the painful sport activity, characterize the type of pain, foot paraesthesias, self-reported ankle instability, and ankle dorsiflexion and eversion muscle power. The Single Assessment Numeric Evaluation (SANE) score will provide a measure of overall leg function.

Adult patients with a confirmed diagnosis of anterolateral CECS, as determined by post-exertional compartment pressure measurements, will be invited to participate in the study. Using concealed, consecutively-numbered randomization envelopes, participants will be randomly assigned to receive either the botulinum (treatment) or the normal saline (control) injection. Participants will answer a web-based outcome questionnaire at Baseline (prior to receiving the injection) and at 2, 4, 6, 8, 12, 16, 24-weeks follow-up. Participants will be asked to do their painful sport activity the day before completing the questionnaire. Ankle dorsiflexion and eversion muscle power will be manually measured by a physiatrist in clinic at 6, 16 and 24-week follow-up visits.

DETAILED DESCRIPTION:
Chronic exertional compartment syndrome (CECS) of the lower leg muscle compartments is a common problem in the active population. The condition often significantly restricts patients from participating in their desired activity to the best of their ability. The pathology of CECS is related to increased intra-muscular pressure related to a restrictive fascia (envelope around the muscle or muscle group). The current standard of care for definitive treatment of CECS is a surgical fasciotomy. However, there have been a number of case reports reporting successful reduction of the symptoms of CECS with intra-muscular botulinum injections. Intra-muscular botulinum injections may reduce the symptoms of CECS by potentially decreasing muscle activation, therefore diminishing blood flow, which may reduce intra-compartmental muscle expansion and pressure of the compartment during exercise. Thus botulinum injections might provide a non-operative method of treating CECS.

This study will determine the effectiveness of intra-muscular botulinum injection, compared to a normal saline placebo, for treatment of lower leg anterolateral CECS, over a 24-week period. Participants will answer a web-based questionnaire before receiving the injection (Baseline) and at regular follow-up intervals at 2, 4, 6, 8, 12, 16, 24-weeks post-injection. The questionnaires will ask the participant to provide detailed information about their painful sport activity, and the maximum level of pain that they experience during that activity. They will also characterize the type of pain experienced, record the time to initial onset and duration of pain during the painful sport activity, and provide an overall measure of their leg function using a Single Assessment Numeric Evaluation (SANE) score. Participants will also attend an in-person appointment in clinic at Baseline, and at 6, 16 and 24-weeks post-injection for assessment of numbness and/or tingling in the foot, ankle instability, and manual ankle muscle power.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of lower leg anterolateral chronic exertional compartment syndrome (CECS), as measured post-exertional compartment pressure measurements of greater than 30 mmHg for immediate post-exertional compartment pressure, and greater than 12 mmHg at 5 minutes after stopping exercise.

Exclusion Criteria:

* Female patients who are pregnant, trying to get pregnant or lactating
* History of keloidal scarring
* History of any significant neurologic disease (ie: amyotrophic lateral sclerosis, motor neuropathy, myasthenia gravis, Lambert-Eaton syndrome)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Change in maximum level of pain at time of painful sport activity from Baseline to 2, 4, 6, 8, 12, 16 and 24-weeks post-injection | Baseline, and 2, 4, 6, 8, 12, 16 and 24-weeks post-injection
  Pain measured on a visual analog scale from 0 to 100, where 0 represents no pain and 100 represents pain as bad as it can be

SECONDARY OUTCOMES:
Change in time to onset of pain during sport activity (minutes) | Baseline, and 2, 4, 6, 8, 12, 16 and 24-weeks post-injection
  Comparison of time to onset of pain during sport activity (minutes) at Baseline to 2, 4, 6, 8, 12, 16 and 24-weeks post-injection
Change in duration of exercise before having to stop due to pain (minutes) | Baseline, and 2, 4, 6, 8, 12, 16 and 24-weeks post-injection
  Comparison of duration of exercise before having to stop due to pain (minutes) at Baseline to 2, 4, 6, 8, 12, 16 and 24-weeks post-injection
Change in duration of pain after stopping painful exercises (minutes) | Baseline, and 2, 4, 6, 8, 12, 16 and 24-weeks post-injection
  Comparison of duration of pain after stopping painful exercises (minutes) at Baseline to 2, 4, 6, 8, 12, 16 and 24-weeks post-injection
Change in the numbness and/or tingling in foot during painful exercises from Baseline to 2, 4, 6, 8, 12, 16 and 24-weeks post-injection | Baseline, and 2, 4, 6, 8, 12, 16 and 24-weeks post-injection
  Presence or absence of numbness and/or tingling in foot during painful exercises
Change in ankle dorsiflexion muscle power from Baseline to 6, 16 and 24-weeks post-injection | Baseline, and 6, 16 and 24-weeks post-injection
  Manual ankle dorsiflexion muscle power test, graded on the following scale:
  0 No muscle activation
  1. Flicker of contraction, but no movement of the ankle joint
  2. Dorsiflexion of the foot with the effect of gravity eliminated
  3. Dorsiflexion of the foot against gravity but no added resistance
  4. Dorsiflexion of the foot against gravity and moderate resistance
  5. Dorsiflexion of the foot against gravity and full resistance
Ankle eversion muscle power | Baseline, and 6, 16 and 24-weeks post-injection
  Manual ankle eversion muscle power test, graded on the following scale:
  0 No muscle activation
  1. Flicker of contraction, but no movement of the ankle joint
  2. Eversion of the foot with the effect of gravity eliminated
  3. Eversion of the foot against gravity but no added resistance
  4. Eversion of the foot against gravity and moderate resistance
  5. Eversion of the foot against gravity and full resistance
Change in Single Assessment Numeric Evaluation (SANE) from Baseline to 2, 4, 6, 8, 12, 16 and 24-weeks post-injection | Baseline, and 2, 4, 6, 8, 12, 16 and 24-weeks post-injection
  Comparison from Baseline to 2, 4, 6, 8, 12, 16 and 24-weeks post-injection for self-assessed rating of overall leg function using a Visual Analog Scale response, where 0 is severely abnormal and 100 is completely normal.
Change in ankle instability from Baseline to 2, 4, 6, 8, 12, 16 and 24-weeks post-injection | Baseline, and 2, 4, 6, 8, 12, 16 and 24-weeks post-injection
  Change in patient-reported assessment of presence or absence of ankle instability from Baseline to 2, 4, 6, 8, 12, 16 and 24-weeks post-injection

CONTACTS AND LOCATIONS:
Overall Officials: Victor Lun, Principal Investigator — University of Calgary Sport Medicine Centre

IPD SHARING:
Plan to Share IPD: No
Requests for individual participant data will be considered upon request.